CLINICAL TRIAL: NCT07345689
Title: A Study to Evaluate the Pharmacokinetics and Safety of Anaprazole Sodium in Subjects With Hepatic or Renal Impairment and in Elderly Subjects
Brief Title: A Study of the Pharmacokinetics and Safety of Anaprazole Sodium in Special Populations
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3571-CPK-1008
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Insufficiency; Renal Insufficiency; Elderly
MeSH Terms: conditions — Hepatic Insufficiency; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy subjects (Experimental): Healthy subjects
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet
- Moderate hepatically impaired subjects (Experimental): Subjects with Child-Pugh B (score 7-9) at the screening visit
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet
- Moderate renal impaired subjects (Experimental): Subjects with eGFR 30-59 mL/min at the screening visit based on the Modification of Diet in Renal Disease (MDRD) equation
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet
- Severe renal impaired subjects (Experimental): Subjects with eGFR 15-29 mL/min at the screening visit based on the MDRD equation
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet
- Elderly subjects (Experimental): Elderly subjects (≥65 years old)
  Interventions: Drug: Anaprazole Sodium enteric-coated tablet

INTERVENTIONS:
Drug: Anaprazole Sodium enteric-coated tablet — 20 mg single dose

SUMMARY:
The objective of this study is to evaluate the pharmacokinetic profile and safety of anaprazole sodium in adult subjects, particularly including the elderly and those with renal or hepatic impairment.

DETAILED DESCRIPTION:
This study is a single-center, open-label, single-dose trial designed to assess the pharmacokinetics and safety of anaprazole sodium in adult subjects. The study consists of five groups: healthy volunteers, subjects with moderate hepatic impairment, subjects with moderate renal impairment, subjects with severe renal impairment, and elderly subjects. Each arm will enroll 8-12 subjects, for a total target sample size of 40-60. The overall trial schedule consists of a Screening Period (Day -14 to Day -2), a Baseline Period (Day -1), a Dosing/Study Period (Day 1 to Day 3), and a Safety Follow-up Period (Day 7). Blood samples for pharmacokinetic (PK) analysis will be collected from all subjects throughout the study. In addition, urine samples for PK assessment will be collected specifically from subjects in the healthy control group and the moderate and severe renal impairment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before any study-related activities commence, demonstrate an understanding of the trial procedures and methodology, and be willing to strictly adhere to the clinical trial protocol for study completion;
2. Subjects (including their partners) must agree to have no plans for conception from screening until 6 months after the last dose of the investigational drug and to voluntarily practice effective contraception during this period;
3. Aged 18 to 70 years (inclusive) at the time of signing informed consent, either male or female. For the elderly group, subjects must be aged 65 years or older (inclusive);
4. Body mass index (BMI) between 18 and 32 kg/m² (inclusive);
5. Subjects in the healthy group should be matched as closely as possible to those in the hepatic impairment, renal impairment, and elderly groups in terms of gender and weight, and additionally matched for age with the hepatic and renal impairment groups;
6. Subjects in the hepatic impairment group must also meet all of the following additional criteria:

   Subjects with chronic liver injury due to primary liver diseases (e.g., hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, etc.), classified as Child-Pugh Grade B hepatic insufficiency; Clinically diagnosed cirrhosis; eGFR > 59 mL/min; Subjects are either those with a stable concomitant medication regimen (for hepatic impairment/complications/other diseases) for ≥2 weeks pre-dose not requiring anticipated adjustment (excluding, e.g., diuretics/insulin), or those not on such medications;
7. Subjects in the renal impairment group must also meet all of the following additional criteria:

Diagnosed with chronic kidney disease (CKD), defined as the presence of any marker of kidney damage or GFR < 60 mL/min for more than 3 months (evidence may include outpatient records, inpatient records, or laboratory reports); GFR must meet the following criteria: Moderate renal impairment (CKD Stage 3): 30-59 mL/min (inclusive); Severe renal impairment (CKD Stage 4): 15-29 mL/min (inclusive); Note: Staging will be determined solely based on the second scheduled GFR measurement during the screening period; Renal function must be stable, defined as meeting either of the following criteria based on two GFR measurements taken prior to dosing (with at least a 3-day interval between measurements): Both results fall within the same CKD stage; or the fluctuation between the two GFR results is <10% (calculated as: [(Second result - First result) / First result] × 100%).

Exclusion Criteria:

1. Subjects with a history of hypersensitivity or allergic constitution (including severe drug allergies or drug hypersensitivity reactions), or with a known allergy to the investigational drug or any of its excipients;
2. QTcF (male) > 470 ms, QTcF (female) > 480 ms;
3. Uncontrolled hypertension, defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg despite antihypertensive therapy. This criterion does not apply to subjects in the healthy group;
4. History of dysphagia or any gastrointestinal disorder that may affect drug absorption, including frequent nausea or vomiting due to any etiology;
5. History of severe infection, trauma, gastrointestinal surgery, or other major surgery within 4 weeks prior to screening;
6. Receipt of any vaccine within 14 days prior to screening, or intention to receive any vaccination during the course of the study;
7. Donation or loss of blood ≥ 400 mL within 3 months prior to screening, or intention to donate blood during the study;
8. Use of moderate or strong CYP3A4 inhibitors/inducers within 2 weeks prior to screening, or planned concomitant use during the study; or use of CYP3A4-sensitive substrates within 2 weeks prior to screening or planned use during the study;
9. Use of proton pump inhibitors (PPIs, e.g., rabeprazole, pantoprazole, esomeprazole) within 2 weeks prior to screening or planned concomitant use during the study; medications known to affect serum creatinine clearance (e.g., calcium dobesilate, trimethoprim/sulfamethoxazole, cimetidine); drugs prone to cause liver injury (e.g., non steroidal anti inflammatory drugs, antibiotics, antituberculosis agents, antifungals, glucocorticoids); or drugs with high plasma protein binding (e.g., warfarin, dicoumarol, diazepam, phenylbutazone, digitoxin);
10. Consumption of special diets (including pitaya, mango, pomelo, and/or xanthine containing foods such as chocolate) within 2 weeks prior to dosing, and/or habitual excessive intake of tea, coffee, grapefruit/grapefruit juice, or caffeinated beverages (average >8 cups per day, 200 mL per cup);
11. History of excessive alcohol consumption, defined as >14 units per week on average, within the 3 months preceding screening (where 1 alcohol unit equals 360 mL of beer, 45 mL of 40% distilled spirits, or 150 mL of wine);
12. Positive result on alcohol breath test or urine drug screening at screening;
13. Average cigarette consumption of ≥10 cigarettes per day within 3 months prior to screening;
14. History of drug abuse or substance misuse;
15. Pregnant or lactating women, or women of childbearing potential with a positive pregnancy test;
16. Intolerance to venipuncture or history of needle/phobia syncope;
17. Use of any investigational drug within 3 months prior to screening or planned participation in another clinical trial during this study;
18. Other conditions deemed by the investigator to compromise the subject's suitability for the study;

    Healthy Subjects will be excluded if they meet any of the following criteria:
19. History of hepatic impairment or renal impairment;
20. Any clinically significant active or chronic disease affecting major organ systems (e.g., circulatory, endocrine, neurological, digestive, respiratory, hematologic, immunologic, psychiatric, or metabolic systems) at screening, or any other medical condition that could potentially confound the interpretation of study outcomes;
21. Clinically significant abnormalities (as judged by the investigator) in physical examination, vital signs, laboratory tests, 12 lead ECG, abdominal ultrasound, or chest X ray;
22. Positive screening result for any of the following: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV antigen/antibody, or syphilis antibody;
23. Administration of any prescription medication, non prescription drug, vitamin supplement, or herbal preparation within 14 days prior to screening;

    Subjects in the hepatic impairment group will be excluded if they meet any of the following criteria:
24. Subjects who present with any of the following conditions and are deemed by the investigator as unsuitable for this study will be excluded:

    Prior liver transplantation; Diseases such as biliary cirrhosis or extrahepatic biliary obstruction;

    Diagnosis of liver cancer or other malignant tumors, with the following exceptions:

    Certain completely cured cancers after surgical resection, such as basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix; Liver cancer patients who have received radical therapy with no recurrence; Liver cancer patients classified as BCLC stage 0. Acute liver failure; History of esophageal or gastric variceal bleeding within 3 months prior to screening;
25. Laboratory test results at screening meeting any of the following criteria:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 × upper limit of normal (ULN);
    2. Absolute neutrophil count < 0.75 × 10⁹/L;
    3. Hemoglobin < 80 g/L;
    4. Alpha fetoprotein (AFP) > 100 ng/mL;
    5. Platelet count < 40 × 10⁹/L; or any other clinically significant laboratory abnormality that, in the investigator's judgment, renders the subject unsuitable for the study;
26. Positive screening result for HIV antigen/antibody; Positive syphilis antibody test result with a confirmatory positive rapid plasma reagin (RPR) test;
27. In addition to the primary hepatic condition, subjects will be excluded if, at screening, they present with any other severe systemic disease-including but not limited to significant gastrointestinal, respiratory, renal, neurologic, hematologic, endocrine, immune, psychiatric, or cardiovascular/cerebrovascular disorders-that in the investigator's judgment would make them unsuitable for the study;

    Subjects in the renal impairment group will be excluded if they meet any of the following criteria:
28. Acute renal failure, prior kidney transplantation, or requirement for renal dialysis during the study;
29. Subjects will be excluded if, in addition to chronic kidney disease and its complications, they have a history or current evidence of any other severe systemic disorder-including but not limited to significant gastrointestinal, respiratory, neurological, hematological, endocrine, oncological (except for completely resected in situ basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, or ductal carcinoma in situ of the breast), immunological, psychiatric, or cardiovascular/cerebrovascular disease-that, in the investigator's opinion, would make participation in the study inappropriate;
30. ALT ≥ 2 × ULN, AST ≥ 2 × ULN; Serum total bilirubin > 1.5 × ULN; Albumin < 30 g/L; Absolute neutrophil count < 1.3 × 10⁹/L; Hemoglobin < 80 g/L; Platelet count < 100 × 10⁹/L; Any other clinically significant laboratory abnormality that, in the investigator's judgment, renders the subject unsuitable for the study;
31. Congestive heart failure classified as New York Heart Association (NYHA) Class III or IV, or Left ventricular ejection fraction (LVEF) < 50% at screening;
32. Positive result for HIV antigen/antibody; Positive syphilis antibody test result, with a confirmatory positive rapid plasma reagin (RPR) test;

    Elderly subjects will be excluded if they meet any of the following criteria:
33. Subjects will be excluded if they have any other severe systemic disease at screening - including but not limited to significant gastrointestinal, respiratory, renal, neurologic, hematologic, endocrine, oncologic (except completely resected in situ basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast), immunologic, psychiatric, or cardiovascular/cerebrovascular disorders - and if, in the investigator's judgment, participation would be inappropriate;
34. Fasting blood glucose > 7.0 mmol/L;
35. ALT ≥ 1.5 × ULN, AST ≥ 1.5 × ULN; Serum total bilirubin > 1.5 × ULN; Albumin < 30 g/L; Creatinine > 1.5 × ULN; Albumin < 30 g/L; Hemoglobin < 100 g/L; Platelet count < 100 × 10⁹/L; Any other clinically significant laboratory abnormality that, in the investigator's judgment, renders the subject unsuitable for the study;
36. Positive screening result for any of the following: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV antigen/antibody, or syphilis antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Up to 48 hours from anaprazole sodium administration
  Cmax of anaprazole sodium in healthy subjects and special participant populations.
Tmax | Up to 48 hours from anaprazole sodium administration
  Tmax of anaprazole sodium in healthy subjects and special participant populations.
AUC0-t | Up to 48 hours from anaprazole sodium administration
  AUC0-t of anaprazole sodium in healthy subjects and special participant populations.
AUC0-∞ | Up to 48 hours from anaprazole sodium administration
  AUC0-∞of anaprazole sodium in healthy subjects and special participant populations.
t1/2 | Up to 48 hours from anaprazole sodium administration
  t1/2 of anaprazole sodium in healthy subjects and special participant populations.
CL/F | Up to 48 hours from anaprazole sodium administration
  CL/F of anaprazole sodium in healthy subjects and special participant populations.
Vz/F | Up to 48 hours from anaprazole sodium administration
  Vz/F of anaprazole sodium in healthy subjects and special participant populations

SECONDARY OUTCOMES:
Number of Subjects With Adverse Events (AEs) | Up to 7 days from the start of administration
  Adverse events are considered to be treatment-emergent if they have started or worsened after first application of study medication to the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, PhD, Principal Investigator — The First Bethune Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China